CLINICAL TRIAL: NCT01300832
Title: The Incidence of Perioperative Deep Venous Thromboses of the Lower Extremities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 10-589-A
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Perioperative DVTs
Keywords: Surgery; Deep Vein Thrombosis; Preoperative
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Duplex scan (Experimental): Subjects undergo preoperative and post-operative duplex scanning of the lower extremities
  Interventions: Procedure: Duplex scan of lower extremities

INTERVENTIONS:
Procedure: Duplex scan of lower extremities — Lower extremities will be duplex scanned pre and post-operatively

SUMMARY:
The study's hypothesis is that there are some patients who come for surgery who have asymptomatic clots in their lower extremities upon their arrival to the hospital for their surgical admission. We will be performing duplex studies of the subjects' legs before their surgery to determine how often clots are present. We will also perform duplex scans of the legs after the subjects' surgeries to determine what factors (surgical, anesthetic, co-morbidities)are correlated with the development of DVTs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ and consentable

Exclusion Criteria:

* Anticoagulation therapy or known DVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The incidence of preoperative DVTs | Day of surgery
Incidence of post-operative DVTs | Within 48 hours of surgery

SECONDARY OUTCOMES:
Risk factors associated with the development of perioperative DVTs | Within 180 days of surgery
Distribution and laterality | Within 180 days of surgery
  Level and laterality of clots that develop and association of these with risk factors
Risks associated with perioperative DVTs | Within 180 days of surgery
  Association of clinical pulmonary emboli and/or cardiac arrests, cerebral vascular events, or other causes of death or significant morbidities (e.g., post-op pneumonias or other infections)perioperatively with DVTs

CONTACTS AND LOCATIONS:
Overall Officials: David Glick, MD, Principal Investigator — University of Illinois at Chicago, Department of Anesthesiology
Locations (1):
- University of Chicago Hospitals, Chicago, Illinois, United States